CLINICAL TRIAL: NCT02791555
Title: Comparison of the Effects of the Direct Thrombin Inhibitor, Pradaxa, to That of Warfarin on Bone Mass and Bone Turnover Markers
Brief Title: Effect of Pradaxa vs Warfarin on Bone Mass and Bone Turnover Markers
Status: Terminated | Type: Observational
Why Stopped: Study was terminated early due to low enrollment numbers.
Sponsor: UConn Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-115-1
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: pradaxa; warfarin
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples w/o DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pradaxa: 20 men and 20 women on Pradaxa for non valvular atrial fibrillation
- Warfarin: 20 men and 20 women on warfarin for non valvular atrial fibrillation, age matched to Pradaxa cohort

SUMMARY:
The investigators are evaluating the effect of Pradaxa in comparison to warfarin on bone turnover and bone density in men and women with atrial fibrillation.

DETAILED DESCRIPTION:
1.0 Hypothesis: The direct thrombin inhibitor Pradaxa positively affects bone turnover markers and increases bone mineral density in women and men at risk for osteoporosis.

2.0 Goal: The goal of this study is to establish if the direct thrombin inhibitor Pradaxa positively affects bone turnover markers and increases bone mineral density in women and men at risk for osteoporosis.

3.0 Specific Aims.

3.1 To determine the effect of Pradaxa on bone mineral density in patients after 6 and 12 months of daily use.

3.2 To determine the effect of the direct thrombin inhibitor Pradaxa on bone turnover markers for osteoclastic resorption (measured as serum levels of C-terminal peptide, and N-telopeptide) and osteoblastic formation (measured as serum levels of bone-specific alkaline phosphatase, osteocalcin and P1NP) in subjects after 6 and 12 months of daily use.

3.3 To evaluate any correlation among the hemoclot, thrombin inhibitor test, changes in markers of bone turnover and changes in bone mineral density in patients on Pradaxa.

3.4 To determine the effect of Pradaxa on change in serum levels of receptor activator of NF B-ligand (RANKL), osteoprotegerin (OPG), RANKL/OPG ratio, inflammatory markers (IL-1b, IL-6, TNF-alpha and FGF-23) and inhibitors of Wnt/beta-catenin signaling pathway including sclerostin and DKK1 at baseline, 6 and 12 months, to understand the mechanisms for the effect of Pradaxa on bone.

4.0 Study design and procedures.

4.1 Study Design:

This will be a prospective, Phase IV age-matched cohort study in men and women who are being started on long-term treatment with Pradaxa for nonvalvular atrial fibrillation. This is a proof of concept study evaluating the effect of Pradaxa, a direct thrombin inhibitor on bone density and bone turnover markers in comparison to warfarin.

4.2 Subject Population:

The investigators will be recruiting patients with nonvalvular atrial fibrillation who are being prescribed Pradaxa by their cardiologists or primary care providers for long-term anticoagulant treatment for participation in the study. The patients taking Pradaxa will be the study group, and will be compared to an age-matched cohort of men and women with nonvalvular atrial fibrillation who are being started on long-term warfarin by their cardiologists or primary care providers (control group). The investigators will be evaluating 20 men and 20 women in the Pradaxa cohort and another age-matched 20 men and 20 women in the warfarin cohort (Pradaxa cohort: N = 40, 20 men, 20 women; Warfarin cohort: N = 40, 20 men, 20 women). The two groups will be determined based on treatment assigned to them by their cardiologists or primary care providers. As age can influence the risk for osteoporosis, the warfarin group will be age-matched to the Pradaxa group for optimal comparison. This will be achieved by offering participation to patients taking warfarin who are similar in age to the patients being recruited for the Pradaxa group. As women are more likely to develop osteoporosis and the effects of Pradaxa may be gender-based as a result of differences in the levels of sex hormones, the investigators are evaluating a cohort of men and women in this pilot study for comparison.

The investigators expect to see an older cohort of subjects with atrial fibrillation, who are also likely to have an increased risk of osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 and above, male and female starting on Pradaxa or Warfarin for nonvalvular atrial fibrillation
2. Able to ambulate independently and travel to UConn Health in Farmington CT-

Exclusion Criteria:

1. Prior known history of osteoporosis
2. Chronic kidney disease with creatinine clearance less than 30
3. Serum 25 hydroxyvitamin D level less than 10
4. Ongoing treatment with medications that interfere with bone metabolism such as steroids, bisphosonates, denosumab, estrogen, SERMS
5. Hypercalcemia, a history of Paget's disease, a history of multiple myeloma, or a history of monoclonal gammopathy of uncertain significance -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female participants age 50 and above with nonvalvular atrial fibrillation being started on Pradaxa or Warfarin
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density in patients | 6 and 12 months
  Measurement of bone density using DXA

SECONDARY OUTCOMES:
Change in bone turnover markers | 6 and 12 months
  Serum C-terminal and N- terminal telopeptide, Bone specific alkaline phosphatase, osteocalcin and P1NP

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lorenzo, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided